CLINICAL TRIAL: NCT00885404
Title: A Prospective, Before and After Study of the Impact of Lower Chloride Intravenous Fluid Management on Patients' Acid-base Status, Renal Profile,Length of Stay and Mortality.
Brief Title: Chloride High Level Of Resuscitation Infusion Chloride High Level Of Resuscitation Infusion Delivered Evaluation
Acronym: CHLORIDE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Austin Health (Other Government)
Responsible Party: Nor'azim Mohd Yunos, Clinical Research Fellow, Department of Intensive Care, Austin Hospital.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2008/03445
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Shock; Critical Illness
Keywords: chloride; acidosis
MeSH Terms: conditions — Shock; Critical Illness; Acidosis | interventions — Ringer's Lactate; Plasmalyte A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous fluids (Other)
  Interventions: Drug: Lower chloride fluids (Hartmann's solution and Plasmalyte®)

INTERVENTIONS:
Drug: Lower chloride fluids (Hartmann's solution and Plasmalyte®) — Intravenous fluids used during the 6 month intervention period (after). Amount of fluids to be used is based on clinicians' discretion.
  Other Names: Plasmalyte; Lactated solution

SUMMARY:
The purpose of this study is to determine whether intravenous fluid management using lower chloride solutions (Hartmann's solutions and Plasmalyte®) will result in better outcome when compared to management using high chloride solutions (0.9% saline and Gelofusine®).

DETAILED DESCRIPTION:
This is a prospective, controlled, before-and-after study. The baseline pre-intervention period will include collection of data while doctors and nurses are unaware that such collection is taking place. During this time, high chloride fluids (saline, Gelofusine, 4% albumin) will continue to be used according to standard practice with an estimated 30,000 liters of saline as well as 2,000 bottles of Gelofusine® being consumed.

Following a wash out period of education and preparation, there will be a complete shift to a working environment where use of saline, Gelofusine and any other fluids with a high chloride level (>110 mmol/L)will be restricted and substituted with fluids of lower chloride concentration similar to blood; either Hartmann's solution or Plasmalyte® or 20% albumin.

The study will compare a 6 month control period (before) and a six month intervention period (after).

ELIGIBILITY:
Inclusion Criteria:

* All Intensive Care Unit (ICU) admissions at Austin Hospital
* All Emergency Department (ED) admissions at Austin Hospital
* All operations at Operating Theatre (OT) with hospital stay of more than 48 hours

Exclusion Criteria: Nil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Mean base excess during hospital stay | Six month control period (before) and 6 month intervention period (after)

SECONDARY OUTCOMES:
Unmeasured anions (strong ion gap) and chloride levels during hospital stay | Six month control period (before) and 6 month intervention period (after)
Serum creatine levels | Six month control period (before) and 6 month intervention period (after)
Length of ICU stay | Six month control period (before) and 6 month intervention period (after)
Length of Emergency Department stay | Six month control period (before) and 6 month intervention period (after)
Length of hospital stay | Six month control period (before) and 6 month intervention period (after)
In-hospital mortality | Six month control period (before) and 6 month intervention period (after)

CONTACTS AND LOCATIONS:
Overall Officials: Nor'azim Mohd Yunos, MBBS, Principal Investigator — Department of Intensive Care, Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Stewart PA. How to understand acid-base. A Quantitative Primer for Biology and Medicine. New York: Elsevier, 1981.
- [Background] Stewart PA. Modern quantitative acid-base chemistry. Can J Physiol Pharmacol. 1983 Dec;61(12):1444-61. doi: 10.1139/y83-207. PMID 6423247
- [Background] Sirker AA, Rhodes A, Grounds RM, Bennett ED. Acid-base physiology: the 'traditional' and the 'modern' approaches. Anaesthesia. 2002 Apr;57(4):348-56. doi: 10.1046/j.0003-2409.2001.02447.x. PMID 11939993
- [Background] Constable PD. Hyperchloremic acidosis: the classic example of strong ion acidosis. Anesth Analg. 2003 Apr;96(4):919-922. doi: 10.1213/01.ANE.0000053256.77500.9D. No abstract available. PMID 12651634
- [Background] Dorje P, Adhikary G, McLaren ID, Bogush S. Dilutional acidosis or altered strong ion difference. Anesthesiology. 1997 Oct;87(4):1011-2; author reply 1013-4. doi: 10.1097/00000542-199710000-00052. No abstract available. PMID 9357917
- [Background] Story DA, Liskaser F, Bellomo R. Saline infusion, acidosis, and the Stewart approach. Anesthesiology. 2000 Feb;92(2):624; author reply 626. doi: 10.1097/00000542-200002000-00053. No abstract available. PMID 10691256
- [Background] Story DA, Poustie S, Bellomo R. Quantitative physical chemistry analysis of acid-base disorders in critically ill patients. Anaesthesia. 2001 Jun;56(6):530-3. doi: 10.1046/j.1365-2044.2001.01983.x. PMID 11412158
- [Background] Reid F, Lobo DN, Williams RN, Rowlands BJ, Allison SP. (Ab)normal saline and physiological Hartmann's solution: a randomized double-blind crossover study. Clin Sci (Lond). 2003 Jan;104(1):17-24. PMID 12519083
- [Background] Dorje P, Adhikary G, Tempe DK. Avoiding latrogenic hyperchloremic acidosis--call for a new crystalloid fluid. Anesthesiology. 2000 Feb;92(2):625-6. doi: 10.1097/00000542-200002000-00055. No abstract available. PMID 10691258
- [Background] Morgan TJ, Venkatesh B, Hall J. Crystalloid strong ion difference determines metabolic acid-base change during in vitro hemodilution. Crit Care Med. 2002 Jan;30(1):157-60. doi: 10.1097/00003246-200201000-00022. PMID 11902256
- [Background] Kellum JA. Fluid resuscitation and hyperchloremic acidosis in experimental sepsis: improved short-term survival and acid-base balance with Hextend compared with saline. Crit Care Med. 2002 Feb;30(2):300-5. doi: 10.1097/00003246-200202000-00006. PMID 11889298
- [Background] Morgan TJ, Venkatesh B, Hall J. Crystalloid strong ion difference determines metabolic acid-base change during acute normovolaemic haemodilution. Intensive Care Med. 2004 Jul;30(7):1432-7. doi: 10.1007/s00134-004-2176-x. Epub 2004 Feb 28. PMID 14991093
- [Background] Story DA, Morimatsu H, Bellomo R. Hyperchloremic acidosis in the critically ill: one of the strong-ion acidoses? Anesth Analg. 2006 Jul;103(1):144-8, table of contents. doi: 10.1213/01.ane.0000221449.67354.52. PMID 16790643
- [Derived] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Derived] Yunos NM, Kim IB, Bellomo R, Bailey M, Ho L, Story D, Gutteridge GA, Hart GK. The biochemical effects of restricting chloride-rich fluids in intensive care. Crit Care Med. 2011 Nov;39(11):2419-24. doi: 10.1097/CCM.0b013e31822571e5. PMID 21705897